CLINICAL TRIAL: NCT01278745
Title: Prevention of Cardiac Allograft Vasculopathy Using Rituximab (Rituxan) Therapy in Cardiac Transplantation (CTOT-11)
Brief Title: Prevention of Cardiac Allograft Vasculopathy Using Rituximab (Rituxan) Therapy in Cardiac Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to inability to meet accrual goals within the funding period
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Clinical Trials in Organ Transplantation (Network); Genentech, Inc. (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAIT CTOT-11
Record Dates: First submitted 2011-01-16; First posted 2011-01-19 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Allograft Vasculopathy; Heart Transplant Recipients
Keywords: cardiac allograft vasculopathy (CAV); prevention; cardiac transplantation; rituximab
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab induction/conventional immunosuppression
  Interventions: Biological: Rituximab induction/conventional immunosuppression (tacrolimus, MMF, and steroid taper)
- Rituximab Placebo (Placebo Comparator): Rituximab Placebo / conventional immunosuppression
  Interventions: Drug: Rituximab placebo/conventional immunosuppression (tacrolimus, MMF, and steroid taper)

INTERVENTIONS:
Biological: Rituximab induction/conventional immunosuppression (tacrolimus, MMF, and steroid taper)
  Arms: Rituximab
Drug: Rituximab placebo/conventional immunosuppression (tacrolimus, MMF, and steroid taper)
  Arms: Rituximab Placebo

SUMMARY:
All people who have a heart transplant are at risk for developing cardiac allograft vasculopathy (CAV). CAV means narrowing of the heart transplant vessels, which is associated with poor heart transplant function. People who develop antibodies after transplant have a higher risk of developing CAV. Infections, high cholesterol, and rejection also increase the risk of developing CAV. People who develop CAV usually have to receive another transplant.

DETAILED DESCRIPTION:
The purpose of this research study is to see if a study drug called rituximab (Rituxan®) prevents CAV. Rituximab destroys certain types of white blood cells called B cells. B cells are important cells in the immune system that help the body fight infection by producing substances called antibodies. B cells and the antibodies they produce are also involved in some kinds of rejection after organ transplantation. Rituximab decreases the number of B cells in the blood and other tissues. The goal of this study is to determine if decreasing B cells with Rituximab can prevent injury to the transplanted heart.

ELIGIBILITY:
Inclusion Criteria for Initial Enrollment:

* Subject must be able to understand and provide informed consent;
* Male or Female, 18 to 75 years of age;
* Candidate for a primary heart transplant (e.g., listed for heart transplant only);
* Historical panel reactive antibodies (PRA) less than 30%;
* Calculated GFR ≥ 40 mL/minute using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI);
* Female and male subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study

Inclusion Criteria for Randomization / Post-transplant:

--Negative PRA within 12 weeks prior to transplant (Local HLA Center Testing) using one of the following:

* One Lambda's LABScreen® Mixed Class I & II (presence or absence), or
* Less than 10% by One Lambda's LABScreen® PRA Class I and II with an MFI of <2000, or
* Calculated panel reactive antibodies (cPRA) less than 10% by LABScreen® Single Antigen testing (Anti-HLA-A, -B, -DR, -DQ). The antigens reported will include those with an MFI >2000.

The Luminex Gen-Probe beads are equivalent to the One Lambda and may be used as an alternative;

* Calculated GFR ≥ 40mL/minute using the CKD-EPI at time of randomization;
* Serum immunoglobulin G (IgG) level greater than 500mg/dL within 90 days prior to randomization;
* Negative test for HIV, HBsAg, HBcAb, and HCV Ab within 12 months prior to transplant. If documentation is not present to support that the testing was performed in the past 12 months, then a blood sample will be collected prior to transplant and sent for local testing. Results may be available after randomization. If positive result, the oversight committee will review the case and provide further recommendations.
* Female subjects of childbearing potential must have a negative pregnancy test.

Exclusion Criteria for Enrollment:

* Prior history of organ transplantation;
* Previous treatment with Rituximab (MabThera® / Rituxan ®);
* Transplant physician intention to use any induction agents;
* History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies;
* History of severe reaction to previous therapy with IVIG;
* Active systemic infection at time of enrollment;
* Any history of serologic positivity to HIV, HBsAg, HBcAb, and HCV Ab;
* History of less than 5 years remission of malignancy. Any history of adequately treated in-situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of the skin will be permitted;
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements;
* Use of other investigational drugs within 4 weeks of enrollment;
* Currently breast-feeding or plans to become pregnant during the timeframe of the study follow-up period.

Exclusion Criteria for Randomization/Post-transplant:

* Recipient of multiple solid organ or tissue transplants;
* Previous treatment with Rituximab (MabThera® / Rituxan ®);
* Use of any induction agents;
* History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies;
* History of severe reaction to previous therapy with IVIG; Lack of IV venous access;
* Active systemic infection at time of randomization;
* Any history of serologic positivity to HIV, HBsAg, HBcAb and HCV Ab;
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements;
* Use of other investigational drugs within 4 weeks prior to randomization;
* Receipt of a live vaccine within 30 days prior to randomization;
* Currently breast-feeding or plans to become pregnant during the timeframe of the study follow-up period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Starling, MD, Study Chair — The Cleveland Clinic; Mohamed Sayegh, MD, Principal Investigator — Brigham and Women's Hospital/Harvard; Anil Chandraker, MD, Study Chair — Brigham and Women's Hospital/Harvard
Locations (24):
- United States (24):
  - Cedars Sinai Heart Institute, Beverly Hills, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Stanford University/Palo Alto VA, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital/CRSTI, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Starling RC, Armstrong B, Bridges ND, Eisen H, Givertz MM, Kfoury AG, Kobashigawa J, Ikle D, Morrison Y, Pinney S, Stehlik J, Tripathi S, Sayegh MH, Chandraker A; CTOT-11 Study Investigators. Accelerated Allograft Vasculopathy With Rituximab After Cardiac Transplantation. J Am Coll Cardiol. 2019 Jul 9;74(1):36-51. doi: 10.1016/j.jacc.2019.04.056. PMID 31272550
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) website — http://www.ctotstudies.org/
- See also: National Heart, Lung, and Blood Institute (NHLBI) website — http://www.nhlbi.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty three out of N=24 participating sites in the United States enrolled 362 participants into this trial. N=163 participants reached the randomization stage of the trial.
Groups:
- Rituximab: Induction: Rituximab was administered in 2 1000 mg doses on Day 0 and Day 12 (+/- 2 days). Maintenance: Mycophenolate Mofetil (MMF) was given at a starting dose of 2-3 g by mouth or intravenously per day in 2 or 3 divided doses. Investigator could choose an alternative treatment if needed. Methylprednisolone/Prednisone dosing was administered according to the local center standard. After 6 months, prednisone was withdrawn at the discretion of the investigator. The suggested oral prednisone taper was Day 14: 20 mg/day by mouth, Day 30: 15 mg/day by mouth, Day 90: 10 mg/day by mouth, Day 180: 5 mg/day by mouth, and greater than Day 180: 0-5 mg/day by mouth. Tacrolimus, was administered per site standards to attain target trough levels. The target whole blood tacrolimus concentrations were as follows: Day 1-30 post transplant 10-20 ng/mL and Day 31-Month 12 5-15 ng/mL.
- Placebo: Induction: Rituximab Placebo was administered in 2 1000 mg doses on Day 0 and Day 12 (+/- 2 days). Maintenance: Mycophenolate Mofetil (MMF) was given at a starting dose of 2-3 g by mouth or intravenously per day in 2 or 3 divided doses. Investigator could choose an alternative treatment if needed. Methylprednisolone/Prednisone dosing was administered according to the local center standard. After 6 months, prednisone was withdrawn at the discretion of the investigator. The suggested oral prednisone taper was Day 14: 20 mg/day by mouth, Day 30: 15 mg/day by mouth, Day 90: 10 mg/day by mouth, Day 180: 5 mg/day by mouth, and greater than Day 180: 0-5 mg/day by mouth. Tacrolimus, was administered per site standards to attain target trough levels. The target whole blood tacrolimus concentrations were as follows: Day 1-30 post transplant 10-20 ng/mL and Day 31-Month 12 5-15 ng/mL.
- Discontinued Pre-Transplant: Subjects that enrolled, but withdrew from the study prior to their transplant.
- Discontinued Pre-Randomization: Subjects that were enrolled and transplanted on study, but withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | Rituximab | Placebo | Discontinued Pre-Transplant | Discontinued Pre-Randomization
Started | 89 | 74 | 121 | 78
Completed | 84 | 68 | 0 | 0
Not Completed | 5 | 6 | 121 | 78
Not completed — Death | 2 | 5 | 7 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 9
Not completed — Withdrawal by Subject | 1 | 1 | 5 | 1
Not completed — Sponsor Decision | 1 | 0 | 62 | 6
Not completed — Ineligible | 0 | 0 | 42 | 61
Not completed — Moves,enrollment in mx studies, et al. | 0 | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 89 | 74 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.80) | 54.8 (11.76) | 54.7 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 73 | 66 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 72 | 62 | 134
  Unknown or Not Reported | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 70 | 57 | 127
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 89 | 74 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Atheroma Volume (PAV)
Description: Nominal or noticeable change, bad or good, from baseline to 1 year in percent atheroma volume (PAV) which is a measure of the degree of coronary arterial obstruction due to host alloimmune processes measured by intravascular ultrasound (IVUS) in a target coronary artery. Thus a decrease in PAV would be an indicator of less obstruction and a better outcome.
Time Frame: Baseline, 1 year
Population: Randomized participants with available data at year one
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 49 | 37
percent | 6.8 (8.21) | 1.9 (4.38)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Test type: Superiority or Other; p = 0.0019, ANCOVA; Adjusted for baseline PAV

2. Secondary Outcome: Death
Description: Participants who died within 12 months post-transplant
Time Frame: 12 months
Population: Randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 3 | 5

3. Secondary Outcome: Re-transplantation or Re-listed for Transplantation
Description: Re-transplantation is defined as the receipt of a subsequent heart transplant and re-listed for transplantation is being listed back on the heart transplant list to be re-transplanted.
Time Frame: 6 to 12 months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 0 | 0

4. Secondary Outcome: Number of Episodes of Biopsy Proven Acute Rejection (BPAR) of Any Grade Per Participant
Description: The number of times a participant experienced biopsy proven acute rejection (BPAR). Biopsy proven acute rejection is when an examination of tissue removed from the transplanted organ indicates that the subject's immune system is trying to reject the graft. BPAR was defined as a biopsy that met the International Society for Heart & Lung Transplantation (ISHLT) criteria to be graded as 1R or greater rejection and was determined by a single, central pathology laboratory.
Time Frame: 6 to 12 months
Population: Randomized participants with at least one centrally read heart biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 86 | 70
Participants
  0 Episodes of BPAR | 45 | 18
  1 Episode of BPAR | 13 | 28
  2 Episodes of BPAR | 17 | 14
  3 Episodes of BPAR | 9 | 8
  4 Episodes of BPAR | 2 | 2

5. Secondary Outcome: Incidence of BPAR (Any Grade)
Description: The number of subjects who experienced any grade of biopsy proven acute rejection (BPAR) within the clinical trial. Biopsy proven acute rejection is when an examination of tissue removed from the transplanted organ indicates that the subject's immune system is trying to reject the graft. BPAR was defined as a biopsy which met The International Society for Heart & Lung Transplantation (ISHLT) criteria to be graded as 1R or greater rejection and was determined by a single, central pathology laboratory.
Time Frame: 6 to 12 months
Population: Randomized participants with at least one centrally read heart biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 86 | 70
Participants | 41 | 52

6. Secondary Outcome: Incidence of AMR
Description: The number of participants who experienced antibody- mediated rejection (AMR). Antibody-mediated rejection (AMR) occurs when the subject develops antibodies directed against the transplanted heart. This was assessed based on local pathology biopsy reads.
Time Frame: 6 to 12 months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 8 | 11

7. Secondary Outcome: Incidence of Cellular Rejection
Description: Cellular Rejection refers to the organ recipient's immune system recognizing a transplanted organ as foreign and mounting a response to it via cellular mechanisms. Cellular rejection was defined as a biopsy which met The International Society for Heart & Lung Transplantation (ISHLT) criteria to be graded as 1R or greater rejection and was determined by a single, central pathology laboratory
Time Frame: 6 to 12 months
Population: Randomized participants with at least one centrally read heart biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 86 | 70
Participants | 41 | 52

8. Secondary Outcome: Incidence of Any Treated Rejection
Description: The number of participants who were treated by their local physician for any type of rejection including, but not limited to cellular rejection and antibody- mediated rejection (AMR) of the transplanted heart regardless of the presence of a biopsy.
Time Frame: 6 to 12 months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 22 | 24

9. Secondary Outcome: Number of Participants With Episodes of Rejection Associated With Hemodynamic Compromise (HDC)
Description: The number of participants that experienced at least one episode of rejection associated with hemodynamic compromise (HDC). Rejection associated with HDC is when there is insufficient blood flow to the transplanted heart in association with acute rejection found in a biopsy. Local biopsies were used for this outcome measure.
Time Frame: 6 to 12 months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 2 | 1

10. Secondary Outcome: Number of Participants With Development of Angiographically Evident Cardiac Allograft Vasculopathy
Description: Cardiac allograft vasculopathy is an aggressive form of atherosclerosis that is characterized by the development of fibrosis affecting cardiac arteries that result in concentric narrowing of the arteries and, ultimately allograft failure. Development of cardiac allograft vasculopathy can be diagnosed via an angiograph which is an X-ray of the cardiac arteries by injecting a radiopaque substance such as iodine.
Time Frame: 1 year
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 19 | 7

11. Secondary Outcome: Number of Participants With Post-transplant Serious Infections Requiring Intravenous Antimicrobial Therapy
Description: Number of participants experiencing at least one serious infection requiring intravenous antimicrobial therapy which is used to kill the growth of microorganisms such as bacteria, fungi, or protozoans.
Time Frame: Transplantation through end of study, up to 1 year post transplantation.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 16 | 13

12. Secondary Outcome: Number of Participants With Post-transplant Incidence of PTLD
Description: The number of participants experiencing at least one post-transplant lymphoproliferative disorder (PTLD) occurrence during this trial. Post-transplant lymphoproliferative disorder is an uncontrolled proliferation of B cell lymphocytes latently infected with Epstein-Barr virus.
Time Frame: Transplantation through end of study, up to 1 year post transplantation.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 0 | 0

13. Secondary Outcome: Post-transplant Safety Outcomes Among Participants: Safety and Tolerability of Rituximab
Description: Defined as participants that experienced at least one adverse event that was possibly, probably, or definitely related to the study drug (i.e., Rituximab or Placebo). Serious adverse events were used to evaluate this endpoint and the attribution was based on the DAIT Medical Monitor's assessment.
Time Frame: Transplantation through end of study, up to 1 year post transplantation
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 89 | 74
Participants | 26 | 26

ADVERSE EVENTS:
Time Frame: From enrollment through end of study (up to one year post randomization)
Arm/Group | Rituximab | Placebo | Discontinued Pre-Transplant | Discontinued Pre-Randomization
Serious Adverse Events (participants affected / at risk) | 55/89 | 45/74 | 0/121 | 1/78
Other Adverse Events (participants affected / at risk) | 29/89 | 26/74 | 0/121 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=89) | Placebo (N=74) | Discontinued Pre-Transplant (N=121) | Discontinued Pre-Randomization (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 10 (10) | 10 (14) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergillosis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocardiosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 6 (6) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complications of transplanted heart (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunosuppressant drug level decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=89) | Placebo (N=74) | Discontinued Pre-Transplant (N=121) | Discontinued Pre-Randomization (N=78)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 7 (7) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 7 (7) | 6 (7) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 4 (4) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 7 (7) | 6 (6) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated with 163 participants randomized, well short of the study's goal of 300 randomized participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No